CLINICAL TRIAL: NCT04829500
Title: Montessori Approaches in Person-Centered Care (MAP-VA): An Effectiveness-Implementation Trial in Community Living Centers
Brief Title: Effectiveness and Implementation of Montessori Approaches in Person-Centered Care Within VA
Acronym: MAP-VA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Center for Applied Research in Dementia (Unknown); University of Alabama at Birmingham (Other); Providence VA Medical Center (U.S. Federal Agency); Edith Nourse Rogers Memorial Veterans Hospital (U.S. Federal Agency); The VA Western New York Healthcare System (U.S. Federal Agency); VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 19-413
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Dementia or a Related Disorder; Mental Health Diagnoses; Symptoms of Agitation or Aggression
Keywords: dementia; mental health; residence characteristics; quality of health care; recreation; long-term care; quality of life
MeSH Terms: conditions — Dementia; Aggression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This 4-year, stepped-wedge cluster randomized trial (SW-CRT) uses a hybrid implementation-effectiveness design, and primary and administrative data collection to pursue four aims. Randomization in this hybrid implementation-effectiveness design is at the system level (in our case the CLC) since existing staff provide the intervention. To address the research questions and corresponding aims, the study approach assesses both the clinical innovation (MAP-VA) and the implementation process itself (blended facilitation). Implementation process measures, fidelity, and outcome indicators will be tracked using a mixed methods evaluation approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-Intervention Baseline Collection Phase (No Intervention): All sites will start with a baseline collection phase without exposure to the intervention, consistent with the stepped wedge cluster randomized trial design. A sequential randomized crossover to the intervention (MAP-VA) will be assigned, which cannot be reversed once it has been introduced.
- MAP-VA Intervention (Experimental): Montessori approaches to person-centered care (MAP-VA) introduces practical strategies that frontline staff can use for successful engagement of residents through retained abilities such as implicit learning, procedural memory, reading abilities. Staff training provides practice with: 1) pre-developed activities and templates, 2) a simple reading assessment to inform development of external cues; and 3) identifying opportunities for increased independence and resident contribution to community routines. Staff are also introduced to concrete strategies that improve dignity, control, and independence.
  Interventions: Behavioral: Montessori Approaches to Person-Centered Care (MAP-VA)

INTERVENTIONS:
Behavioral: Montessori Approaches to Person-Centered Care (MAP-VA) — Montessori approaches to person-centered care (MAP-VA) introduces practical strategies that frontline staff can use for successful engagement of residents through retained abilities. Staff are also introduced to concrete strategies that improve dignity, control, and independence. MAP-VA is based on the work of Maria Montessori who demonstrated that a structured, supportive environment and meaningful, active roles in the classroom enabled children to fulfill their greatest potential physically, mentally, and emotionally. Montessori principles have been applied to dementia care for more than 20 years to promote functional independence, meaningful engagement, and dignity.
  Other Names: Montessori Activity Programming, Montessori Inspired Lifestyle, Montessori for Dementia
  Arms: MAP-VA Intervention

SUMMARY:
Background: Addressing behavioral and neuropsychiatric symptoms of Veterans with dementia and serious mental illness (SMI) such as schizophrenia can be challenging for staff in VA long-term care settings, called Community Living Centers or CLCs. These behaviors of distress (agitation, aggression, and mood disturbance) are not just associated with staff stress and burnout; they also hasten residents' functional decline, decrease quality of life, and increase mortality. Staff training in non-pharmacological interventions can be effective. Yet systems barriers, task-based care models, and time constraints often result in staff employing "quicker," less effective strategies. Montessori Approaches to Person-Centered Care for VA (MAP-VA)- a staff training, intervention, and delivery toolkit- developed in collaboration with VA operational partners, Veterans, and frontline CLC staff is positioned to respond to this challenge. The investigators' prior work shows probable impacts on CLC quality indicators at the individual and unit level (e.g., psychotropic medications, depressive symptoms, weight loss, falls, pain). The goal of this study is to evaluate the MAP-VA program and necessary supports for a successful implementation at 8 VA CLCs.

Significance/ Innovation: VHA's Modernization Plan focuses on empowering front-line staff to lead quality improvement efforts like the ones taught through MAP-VA. MAP-VA is distinct from existing interventions in its: 1) application to Veterans with a range of diagnoses and cognitive abilities; 2) emphasis on pairing practical skill-building for staff with overcoming system-level barriers that inhibit person-centered care; and 3) engagement of all staff rather than a reliance on provider-level champions. Yet, MAP-VA is a complex intervention that requires participation of multiple stakeholder groups, making implementation facilitation necessary. To date, no studies have evaluated MAP implementation success in operational settings (community or VA) and sustainability is rarely examined.

Aims: This 4-year study will examine both the effectiveness of the MAP-VA program on resident outcomes, person-centered care practices, and organizational culture as well as an evaluation of the implementation barriers to adopting MAP-VA in a sustainable way over a 12 month period. Staff and residents at 8 CLCs will participate in the study.

DETAILED DESCRIPTION:
Specific Aims: A hybrid implementation-effectiveness study is necessary to evaluate MAP-VA for Veterans and staff in CLCs. Study Aims include: 1) evaluate implementation facilitation and identify barriers to MAP-VA adoption and fidelity; 2) determine effectiveness of MAP-VA implementation on resident behavioral, emotional, and physical health outcomes; 3) determine effectiveness of MAP-VA implementation on person-centered care practices and organizational culture; and 4) examine the extent to which MAP-VA is sustained after external facilitation support has ended.

Methodology: A stepped-wedge cluster randomized controlled trial will be used to evaluate within- and between-cluster implementation success and treatment effects over 18 months. Eight CLCs (approximately 24 CLC neighborhoods) will be randomized to a sequential crossover to the intervention with six months of facilitation. Sequential balancing will be used during randomization to balance the sample over time. Analyses will account for time trends and correlations within cluster. Normalization process theory and the RE-AIM evaluation framework will guide the implementation evaluation and integration of qualitative and quantitative data. Data sources include primary data collection (e.g., resident interviews, staff interviews, surveys, researcher observation) and existing VA administrative data (e.g., Minimum Data Set 3.0, pharmacy, annual employee survey).

The unit of analysis in hybrid implementation-effectiveness designs is typically at the system level (in the investigators' case the CLC/neighborhood) since existing staff provide the intervention. To address the research questions and corresponding aims, the study approach assesses both the clinical innovation (MAP-VA) and the implementation process itself (Blended Facilitation). Implementation process measures, fidelity, and outcome indicators will be tracked using a mixed methods evaluation approach. Common features of SW-CRTs utilized in this study include: 1) a baseline collection phase where no clusters are exposed to the intervention; 2) sequential randomized crossover to the intervention (MAP-VA), which cannot be reversed once it has been introduced; and 3) analyses that account for time trends and correlations within clusters. Randomization of facilities to MAP-VA will simply delay its rollout to sites randomized later in the sequence (like a wait-list control condition).

Target sample size and analyses. A sample size of more than 200 CLC Staff and 96 Veteran residents are anticipated. Qualitative interview data will be analyzed using a content analytic approach. To test Aims 2 and 3 (effectiveness of MAP-VA) on the primary effectiveness outcome, scores for residents in the pre-intervention control condition will be compared to scores from residents in the intervention condition. GEE models with an identity link will be used to examine and compare means over time, with time considered a random effect. An indicator term will denote if the observation is pre- or post- intervention implementation, thus representing whether there was an overall difference during the intervention period versus the pre-intervention period.

A centralized Data Safety Monitoring Board coordinated through the study sponsor (VA Health Services R&D) will convene to review study materials annually.

ELIGIBILITY:
Inclusion Criteria:

Residents who meet at least one of the following eligibility criteria will be eligible:

* dementia diagnosis or related disorder
* Cognitive Function Scale score indicative of impairment
* positive Patient Health Questionnaire (PHQ-9) depression score
* mental health diagnosis (e.g., ICD-10 codes)
* indication of agitation or aggression per MDS behavior items
* active prescription for a PRN or scheduled antipsychotic, sedative/hypnotic, or benzodiazepine/anxiolytic

Exclusion Criteria:

* Residents admitted for hospice or respite care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in resident agitation from pre-intervention to post-intervention | Primary data collection occurs at 4 time points across 7 months (2 pre-intervention and 2 after the intervention has been initiated)
  Staff-reported observations of resident agitation will be collected over time using the Cohen-Mansfield Agitation Inventory (CMAI). The CMAI is a widely used, valid measure of agitation frequency for older adults across diagnoses in NH settings. Staff rate 29 behaviors over the past two weeks (1=never to 7=several times/hr) across four subscales: verbally nonaggressive behaviors, verbally aggressive behaviors, physically nonaggressive behaviors, and physically aggressive behaviors. Higher scores indicate more agitation.

SECONDARY OUTCOMES:
Change in resident mood from pre-intervention to post-intervention | Primary data collection occurs at 4 time points across 7 months (2 pre-intervention and 2 after the intervention has been initiated)
  Resident symptoms of depression will be assessed using the 9-item Patient Health Questionnaire (PHQ-9) or the PHQ-Observational (PHQ-OV) for residents who cannot self-report mood symptoms. Staff or residents will be asked to rate the frequency of symptoms over the past 2 weeks on a 4-point scale (0 = never or 1 day, to 3 = nearly every day). Higher scores indicate more mood symptoms.
Change in resident psychotropic medication use from pre-intervention to post-intervention | Monthly pharmacy data will be examined pre-and post-intervention for time trends.
  Psychotropic medication use will be extracted for individual residents enrolled in the study as well as examined at the unit-level using pharmacy data. Monthly administration rates of PRN anti-psychotics, benzodiazepines, and sedatives / hypnotics often used for agitation will be tracked.
Change in patient-centered care practices / organizational culture from pre-intervention to post-intervention | Primary data collection occurs at 4 time points across 7 months (2 pre-intervention and 2 after the intervention has been initiated)
  Staff-rated patient-centered care practices (e.g., atmosphere, individualized care and services) will be assessed using subscales of the Patient Centered Care Practices in Assisted Living (PC-PAL). Items are rated on a 4-point scale from 1 = strongly disagree to 4 = strongly agree, with higher scores indicating higher patient-centered care practices.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Marie Hilgeman, PhD, Principal Investigator — Tuscaloosa VA Medical Center, Tuscaloosa, AL
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created at the end of the study. The study team does not have access to a data repository infrastructure; therefore specific requests for use of the final data will be considered by contacting the local team.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after all primary manuscripts and reports have been completed after study closure.

REFERENCES:
- [Result] Kennedy KA, Snow AL, Mills WL, Haigh S, Mochel A, Curyto K, Bishop T, Hartmann CW, Camp CJ, Hilgeman MM. Implementing Montessori approaches after training: A mixed methods study to examine staff understanding and movement toward action. Dementia (London). 2024 Oct;23(7):1126-1151. doi: 10.1177/14713012241263712. Epub 2024 Jul 22. PMID 39039035

DOCUMENTS (1):
  • Informed Consent Form (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT04829500/ICF_000.pdf